CLINICAL TRIAL: NCT06898866
Title: An Effectiveness-Implementation Trial of Functional Restoration for Chronic Pain Management in Active Duty Military Personnel
Brief Title: Functional and Occupational Rehabilitation of Troops
Acronym: FORT
Status: Not yet recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00001264; W81XWH-22-2-0041 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-03-18; First posted 2025-03-27 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Chronic Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Treatment as Usual: At their assigned step, each site will receive 6 months of Treatment as Usual (TAU). This step will include patients seen at each of the six study sites who participate in the current interdisciplinary chronic pain management program that is available at those sites prior to the initiation of the FORT Implementation Facilitation.
- Implementation Facilitation + FORT: At their assigned step, each site will receive 6 months of External Facilitation kicked off with an initial site visit. At the site visit, the external facilitators will meet with key stakeholders, clinic providers, and staff. Together, the team will review the FORT Implementation Site-Assessment Survey as a baseline assessment of implementation as well as the FORT Program Implementation Planning Guide. The team will work together to develop a site-specific implementation blueprint called the Site Action Plan.
- FORT Functional Restoration: During the subsequent 6 months, the site action plan will be executed, monitored, and refined to meet the implementation goals. As per Implementation Facilitation, the facilitator will apply many different implementation strategies to support the uptake of FORT, tailoring strategies to the needs of the site and the stakeholders engaged in the process. Implementation Facilitation will be conducted virtually through a combination of scheduled video teleconferences or phone calls. Regular implementation team meetings will be scheduled to support the implementation process

SUMMARY:
The proposed implementation science project will evaluate the factors that support or hinder the successful implementation of the FORT Functional Restoration Program at six Military Treatment Facilities (MTF) across the Military Health System. It will also evaluate the associated effectiveness outcomes related to chronic musculoskeletal pain management in active-duty military personnel.

DETAILED DESCRIPTION:
This project will be an effectiveness-implementation hybrid type 2 study design using a stepped-wedge randomized clinical trial research design. The study will simultaneously evaluate clinical and implementation outcomes related to the establishment of functional restoration programs. The study investigators have collaborated with the Defense Health Agency (DHA) Pain Management Clinical Support Services to identify chronic pain management programs at six MTFs interested in systematically improving and assessing the outcomes of their program. The MTFs will be randomized in pairs to initiate the Implementation Facilitation strategy to improve the implementation of their program over three 6-month intervals, after an initial 6-month baseline. This hybrid design will allow for the evaluation of both implementation and clinical effectiveness research aims and support rapid translation of research outcomes. Each site will participate in a minimum 6-month baseline period prior to the intervention period to serve as its own treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

"patient referred to functional restoration program by provider"

Exclusion Criteria:

"patient not referred to functional restoration program by provider"

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Active duty military personnel diagnosed with chronic musculoskeletal pain.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Pain Impact Score (PIS) | Baseline to 13 months
  The Pain Impact Score (PIS) is based on the Defense and Veterans Pain Rating Scale (DVPRS), which measures 7-day average pain intensity (0-10 scale) and adaptive PROMIS pain interference and physical function using numeric, color, facial, and word descriptors and is validated. PROMIS T-scores are converted to compute the PIS, ranging from 8-50 with a higher score indicating greater pain.

IPD SHARING:
Plan to Share IPD: Undecided